CLINICAL TRIAL: NCT02858050
Title: A Randomized, Parallel-group, Pilot Study on the Effect of Using the Portal724-Medication Electronic Medication System (MEMS) Smart Cap With Real-time Medication Adherence Among Patients Being Treated With Grazoprevir/Elbasvir
Brief Title: Portal-724 MEMS for Medication Adherence Patients Taking HCV Medications
Status: Completed | Type: Observational
Sponsor: Saint Michael's Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jihad Slim, MD, Chief and Program Director, Infectious Diseases, Saint Michael's Medical Center
Other Study IDs: 13/16
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MEMs Cap Real-Time Monitoring: Group 1 will consist of patient taking hepatitis C medicaitons and will have Portal-724 MEMs cap place in their medication bottle and will transmit data in real-time
  Interventions: Device: Portal-724 MEMs Cap
- MEMs Cap Without Real-Time Monitoring: Group 2 will consist of patient taking hepatitis C medicaitons and will have Portal-724 MEMs cap place in their medication bottle and data will be downloaded at each study visit while taking hepatitis C medications
  Interventions: Device: Portal-724 MEMs Cap

INTERVENTIONS:
Device: Portal-724 MEMs Cap

SUMMARY:
The study will look at real-time adherence monitoring with Portal-724 MEMS cap. It integrates medication bottle, Smart Cap, Pill Dispenser, Embedded Computer, Embedded Cellular Modem and Tamper Proof apparatus. This device is capable of transmitting pill dispensing events from the patient's home to the Cloud over Cellular and IP networks. The transmission is done in real time if cellular coverage is above 1-bar, but if the cell signal is not available or if the signal is below the threshold, then the device Store-and-Forward feature is automatically activated. The patient will be randomized to real-time monitoring or to have monitoring data download monthly at each study visit while taking hepatitis C medications

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a very important health problem worldwide. Majority of the estimated 160 million people infected globally are unaware of their affliction [1]. It is a leading cause of chronic hepatitis, liver cirrhosis, and hepatocellular carcinoma. In the United States alone, HCV infection is the most common chronic blood-borne infection, affecting about 3.2 million individuals The study will look at real-time adherence monitoring with Portal-724 MEMS cap. It integrates medication bottle, Smart Cap, Pill Dispenser, Embedded Computer, Embedded Cellular Modem and Tamper Proof apparatus. This device is capable of transmitting pill dispensing events from the patient's home to the Cloud over Cellular and IP networks. The transmission is done in real time if cellular coverage is above 1-bar, but if the cell signal is not available or if the signal is below the threshold, then the device Store-and-Forward feature is automatically activated. The patient will be randomized to real-time monitoring or to have monitoring data download monthly at each study visit while taking hepatitis C medications

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years old and above.
2. HCV treatment naïve or HCV trreatment experienced
3. HCV RNA PCR > 10,000 IU/L
4. Confirmed infection with Hepatitis C virus (HCV) by HCV serum antibody assay and by HCV Ribonucleic Acid (RNA) Polymerase Chain Reaction (PCR) and Confirmed chronicity with 2 PCR's 6 months apart.
5. Patients with HCV Genotype 1, 4
6. Patients are candidates for treatment of HCV with oral Direct-Acting Agents (DAA)
7. understand the study procedures, alternative treatments available, risks involved with the study, and voluntarily agrees to participate by giving written informed consent

Exclusion Criteria:

1. Patient not willing to sign written informed consent
2. Patients deemed not suitable for HCV treatment as deemed by the treating physician at the liver center
3. Patients with decompensated liver cirrhosis, defined as follows:

   1. Liver biopsy within the last year showing Scheuer Stage 4 or transient elastography (Fibroscan®) in the last year with a reading of >12.5 kPa; AND
   2. Any clinical sign of hepatic decompensation such as ascites (fluid in the abdomen), jaundice (yellowing of eyes and skin), esophageal varices with bleeding (enlarged veins of the esophagus seen on endoscopy) or hepatic encephalopathy (tremors, confusion, sleepiness)
4. Co-Infection with the Hepatitis B virus
5. Any liver disease of non-HCV etiology such as Hemochromatosis, Wilson's Disease, Alcoholic liver disease or Non-Alcoholic Steato-Hepatitis (NASH)
6. Hepatocellular carcinoma or any other malignancy
7. Untreated psychiatric conditions such as major depression, schizophrenia, bipolar disorder which in the opinion of the Principal Investigator will not interfere with protocol visit and/or procedures
8. Current and untreated substance abuse (cocaine, opiates, alcohol, marijuana, other recreational drugs, controlled substances)
9. Patient is pregnant or breastfeeding.
10. Patients unwilling to use cellular phones
11. Patients unwilling to follow specific instructions for medication intake
12. Patient has any of the following conditions:

    * Organ transplants (including hematopoietic stem cell transplants) other than cornea and hair.
    * Poor venous access that precludes routine peripheral blood sampling required for this trial.
    * History of gastric surgery (e.g., stapling, bypass) or subject with a history of malabsorption disorders (e.g., celiac sprue disease).
    * History of a medical/surgical condition that resulted in hospitalization within the 3 months prior to enrollment, other than for minor elective procedures
    * Medical/surgical conditions that may result in a need for hospitalization during the period of the study
    * any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, TNF antagonists, or other immunosuppressant drugs during the course of the trial
13. has exclusionary laboratory values as listed below: Noncirrhotic/Cirrhotic Subjects Creatinine clearance < 50 mL/min Hemoglobin <9.5 g/dL for both male and female subjects Platelets <50 x 103/μL serum albumin < 3.0 g/dL INR >1.7, unless subject has a stable INR on an anticoagulant regimen. HbA1c >10% ALT >10XULN AST >10XULN
14. is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve and treatment-experienced genotype 1 or 4 HCV patients with or without compensated cirrhosis will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Slim, MD, Principal Investigator — Saint Micahel's Medical Center
Locations (1):
- Saint Michael's Medical Center, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Portal-724 MEMs Cap Real-Time Monitoring: Group 1 will consist of patient taking hepatitis C medicaitons and will have Portal-724 MEMs cap place in their medication bottle and will transmit data in real-time
  Portal-724 MEMs Cap
- Portal-724 MEMs Cap Without Real-Time Monitoring: Group 2 will consist of patient taking hepatitis C medicaitons and will have Portal-724 MEMs cap place in their medication bottle and data will be downloaded at each study visit while taking hepatitis C medications
  Portal-724 MEMs Cap
Period: Overall Study
Arm/Group | Portal-724 MEMs Cap Real-Time Monitoring | Portal-724 MEMs Cap Without Real-Time Monitoring
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portal-724 MEMs Cap Real-Time Monitoring | Portal-724 MEMs Cap Without Real-Time Monitoring | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 12 | 14 | 26
  Race: Non-Caucasion | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Treatment Naive [Count of Participants; unit: Participants] | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Use of Portal724-MEMS Service on Medication Adherence in the Treatment of Hepatitis C in Patients, Defined as Compliance to Regimen 95% of the Time.
Description: Number of Participants with Compliance to Regimen 95% of the Time Due to Portal724-MEMS Service
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Portal-724 MEMs Cap Real-Time Monitoring | Portal-724 MEMs Cap Without Real-Time Monitoring
Number analyzed (Participants) | 20 | 20
Participants | 19 | 18
Statistical Analysis 1: Comparison: Portal-724 MEMs Cap Real-Time Monitoring vs Portal-724 MEMs Cap Without Real-Time Monitoring; Test type: Other; p = 0.548306, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Portal-724 MEMs Cap Real-Time Monitoring | Portal-724 MEMs Cap Without Real-Time Monitoring
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
A limitation to our pilot study might be the small sample size and a larger study might detect a difference in adherence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT02858050/Prot_SAP_000.pdf